CLINICAL TRIAL: NCT05575141
Title: Robotic Versus Open Comparison in the Surgical Treatment of Wide Abdominal Wall Hernias: a Multicenter International Randomized Controlled Trial
Brief Title: Robotic Versus Open Comparison in the Surgical Treatment of Wide Abdominal Wall heRnias (ROCSTAR)
Acronym: ROCSTAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Head of General Surgery, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROCSTAR
Record Dates: First submitted 2022-04-02; First posted 2022-10-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Ventral Incisional Hernia; Abdominal Wall Hernia
Keywords: Abdominal Wall Hernia; robotic TAR (rTAR); open TAR (oTAR); transversus abdominis release (TAR)
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Intervention Model Description: a multicenter international randomized controlled trial
Masking Description: This is an open-label Randomized Controlled Trial (RCT) where the patient, surgeon, research coordinators and hospital staff will be aware of the treatment arm after randomization. As the open approach is performed using a large midline incision, whereas the robotic approach applies only 6 or 7 small incisions (or less if no posterior component separation is needed), blinding of patients and physicians is difficult.
  Evaluation of the radiographic imaging of the abdominal wall at 24 months (MRI or CT scan) will be done by radiologists at the local participating center blinded to the randomized treatment arm. This will be a blinded evaluation for the presence or absence of hernia recurrence. Data analysis will be performed in a blinded manner by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTAR (Active Comparator): Patients randomized in the robotic group will undergo the technique for intra-and perioperative management for robotic complex abdominal wall repair cases as used in the center. A robotic surgical platform (da Vinci X or da Vinci Xi Surgical System, Intuitive Surgical, Aubonne, Switzerland) will be used and a retrorectus +/- retromuscular mesh placement performed. Use of component separation or not will be at the discretion of the surgeon. In principle the posterior layer and the anterior fascia will be closed avoiding a bridging technique. Drain management and mesh fixation are left to the surgeon's preference.
  Interventions: Procedure: incisional hernia repair
- oTAR (Active Comparator): Patients randomized in the open group will undergo the technique for intra-and perioperative management for open complex abdominal wall repair cases as used in the center. A retrorectus +/- retromuscular mesh placement performed. Use of component separation or not will be at the discretion of the surgeon. In principle the posterior layer and the anterior fascia will be closed avoiding a bridging technique. Drain management and mesh fixation are left to the surgeon's preference.
  Interventions: Procedure: incisional hernia repair

INTERVENTIONS:
Procedure: incisional hernia repair — Incisional hernia repair for the treatment of wide ventral incisional hernias.

SUMMARY:
In the treatment of ventral incisional hernias, a mesh repair in the retromuscular plane is considered as the gold standard. To allow for adequate medialization of the fascial borders and a complete closure of the defect in case of large incisional hernias, component separation techniques are increasingly being used. When compared to anterior component separation, posterior component separation by transversus abdominis release (TAR) seems to decrease postoperative wound problems. While laparoscopic techniques pose significant difficulties to perform TAR minimally invasively (mainly due to ergonomic and technical reasons), these limitations seem to be overcome by robotic platforms. Initial retrospective patient series report on significantly shorter postoperative hospital stay and fewer complications after robotic transversus abdominis release (rTAR), when compared to open transversus abdominis release (oTAR). High-quality prospective evidence on rTAR is currently lacking.

ELIGIBILITY:
Inclusion Criteria:

- All patients requiring treatment of a wide ventral incisional hernia (of more than 8 centimetres in width)

Exclusion Criteria:

* Pregnant or suspected pregnancy
* Not-curatively treated malignancy, with life expectancy less than 24 months
* Patients unable to give informed consent or complete study specific questionnaires
* Emergency surgery
* Primary ventral hernia repair
* Exclusively lateral hernias not involving the midline
* Incisional hernia repair after open abdomen or enterocutaneous fistula
* Active wound infection
* Previous anterior or posterior component separation
* Patients with an existing ostomy
* Patients with a life expectancy of less than 24 months
* Patients suspected of being unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | hours from the end of surgery (last skin suture) until discharge, assessed up to 20 days
  Length of postoperative hospital stay

SECONDARY OUTCOMES:
Skin-to-skin operative time | Per-operative (minutes)
  Skin-to-skin operative time from first incision until last skin suture
Conversion rate | Per-operative
  Conversion rate from the robotic-assisted approach to the open approach
Surgical site related complications | 30 days
  Surgical site infection - surgical site occurrence - surgical site occurrence requiring procedural interventions
Readmission rate | 30 Days and 3 months postoperative
  Readmission rate
Post-anesthetic discharge scoring system | From the end of surgery (last skin suture) until discharge, assessed up to 20 days
  Minimum score is 0, maximum score is 12. The higher the score, the better the outcome.
Postoperative visual analogue scale pain score | From the end of surgery (last skin suture) until discharge, assessed up to 20 days
  Minimum score is 0, maximum score is 10. The higher the score, the worse the outcome.
EuraHS Quality of Life Scoring | Preoperatively, 30 days, 3 months, 12 months, 24 months, 60 months
  Minimum score is 0, maximum score is 90. The higher the score, the worse the outcome.
Body Image Scale | Preoperatively, 30 days, 3 months, 12 months, 24 months, 60 months
  Minimum score is 0, maximum score is 10. A higher score means a higher level of body image disturbance (worse outcome).
Hernia recurrence | 30 days, 3 Months, 12 months, 24 months, 60 months
  Hernia recurrence
Reoperation for hernia recurrence or abdominal surgery not for hernia recurrence | 30 days, 3 Months, 12 months, 24 months, 60 months
  Reoperation for hernia recurrence or abdominal surgery not for hernia recurrence
Postoperative complications | 30 days
  Postoperative complications classified acoording to the Clavien-Dindo Classification
Reoperation rate | 30 days
  Reoperation rate

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD PhD, Principal Investigator — Clinical research center Maria Middelares

IPD SHARING:
Plan to Share IPD: No